CLINICAL TRIAL: NCT07055581
Title: A Phase II Study of Durvalumab Combined With EP Prior to Chemoradiotherapy and Followed by Durvalumab as Consolidation for Patients With Limited-stage Small-cell Lung Cancer (CONCUR Study)
Brief Title: Durvalumab as Consolidation for Patients LS-SCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qian Chu (Other)
Responsible Party: Sponsor-Investigator, Qian Chu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-24-22526
Record Dates: First submitted 2025-06-17; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer Limited Stage
Keywords: small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- single arm, multi-center, phase II study (Experimental)
  Interventions: Drug: Induction Durvalumab +etoposide/platinum +Radiochemotherapy+ durvalumab maintenance

INTERVENTIONS:
Drug: Induction Durvalumab +etoposide/platinum +Radiochemotherapy+ durvalumab maintenance — Drug: Durvalumab
  Induction Phase: Durvalumab (1500mg D1 IV Q3W) combined with EP [cisplatin or alternatively Carboplatin (AUC 5-6 D1) and Etoposide (100 mg/m² (BSA) D1-3) once every 3 weeks] for minimum two cycles prior to thoracic radiotherapy Consolidation Phase: Durvalumab (1500 mg once every 4 weeks) until PD or unacceptable toxicities or for a maximum of 24 months, whichever occurs first.
  Drug: Chemotherapy Concomitant chemoradiotherapy consists of further four cycles Etoposide (100 mg/m² D1-3), cisplatin (75 mg/m² D1) /carboplatin (AUC 5-6 D1) q3w
  Radiation: Thoracic Radiotherapy Radiotherapy to the primary tumor is recommended to start with the 3rd cycle of EP, which can be delayed appropriately per investigator's decision. 60±6 Gy, 1.8-2 Gy/d or 45±1.5 Gy (1.5 Gy per fraction twice daily, with 4 hours or more between fractions) or other biologically equivalent regimens will be delivered.

SUMMARY:
Small-Cell Lung Cancer (SCLC) accounts for 10% to 15% of new lung cancers and is a highly aggressive neuroendocrine tumor. In the past 30 years, the treatment of SCLC has made very limited progress, and basically made breakthroughs in radiotherapy and chemotherapy. With the advent of the immune era, immunotherapy has achieved initial results in the treatment of SCLC. Approximately one-third of patients with small cell lung cancer are in limited-stage (LS-SCLC) disease at first diagnosis. Except for a very small number of patients with T1-2N0 who can be treated with surgery or stereotactic radiation therapy (SBRT), the standard treatment for the rest of the patients with LS-SCLC is concurrent chemoradiotherapy. The ORR of platinum-combined etoposide regimen combined with thoracic radiotherapy in LS-SCLC can reach 70% to 90%, and the median OS is 16-24 months, which significantly improves the survival of patients. Although many measures have been taken in the treatment of LS-SCLC, only 20% of LS-SCLC can be cured, and most patients have relapse and metastasis after treatment. This study is a single arm phase II preliminary pilot study, aim to assess the efficacy and safety of durvalumab combined with EP prior to CRT and followed by durvalumab consolidation therapy for LS-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1.Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* 2.Histologically or cytologically confirmed small cell lung cancer
* 3.Limited-stage, defined as stage I-III SCLC (T any, N any, M0). Patients who are Stage I or II must be medically inoperable as determined by investigator.
* 4.Age > 18 years.
* 5.Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* 6.Adequate normal organ and marrow function.
* 7.Must have a life expectancy of at least 12 week.
* 8.At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to enrollment.

Exclusion Criteria:

* 1.Patients with extensive disease small-cell lung cancer.
* 2.Patients who previously received radiotherapy to the thorax or chemotherapy for small cell lung cancer.
* 3.Any previous diagnosis of transformed non-small cell lung cancer (NSCLC), epidermal growth factor receptor (EGFR) activating mutation positive NSCLC that has transformed to SCLC, or mixed SCLC NSCLC histology. Patients with mixed histology tumors with predominant SCLC histology are allowed.
* 4.Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values.
* 5.Any concurrent chemotherapy other than study treatment, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* 6.History of allogenic organ transplantation.
* 7.Active or prior documented autoimmune or inflammatory disorders.
* 8.Uncontrolled intercurrent illness.
* 9.History of leptomeningeal carcinomatosis.
* 10.Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
* 11.History of active primary immunodeficiency
* 12.Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of antiHBc and absence of HBsAg) and with undetectable HBV DNA (< 10 IU/ml or under the limit of detection per local lab standard) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* 13.Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
* 14.Prior treatment in a previous durvalumab clinical study.
* 15.Known allergy or hypersensitivity to IP or any excipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Every 6weeks from the beginning of Cycle 1(each cycle is 42±7days) in induction phase, every 8weeks(each cycle is 56±7days) in first year and every 12weeks in second year in consolidation phase, thereafter every 24weeks until PD or death,up to 3years
  Defined as the time from first dose of study treatment to date of the first objective disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 3 years after the first patient was enrolled. OS rate at 1 year(%), 2 years(%) and 3 years(%) are presented.
  Defined as the time from first dose of study treatment to date of death from any cause.
Objective response rate (ORR) | up to 3 years
  Defined as the percentage of patients with at least 1 assessment result of complete response (CR) or partial response (PR) based on all enrolled patients with evaluable disease per RECIST 1.1.
DoR （Duration of response） | From the date of first documented response until the first date of documented progression or death in the absence of disease progression ,up to 3 years
  Defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression (i.e. date of PFS event or censoring - date of first response +1).
Number and proportion of patients with adverse events | Approximately 3 years
  AE, SAE, AESI, TRAE, imAE will be recorded by Common Terminology Criteria of Adverse Events version 5 [CTCAE v.5],number and proportion of patients will be described.

IPD SHARING:
Plan to Share IPD: No